CLINICAL TRIAL: NCT05213949
Title: An Observational Study of Risk Factors and Long-term Prognosis of Patients With Pyogenic Liver Abscess in the "Real-world"
Brief Title: An Observational Study of Risk Factors and Long-term Prognosis of Patients With Liver Abscess in the "Real-world"
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2021-355
Record Dates: First submitted 2021-12-30; First posted 2022-01-28 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Liver Abscess, Pyogenic; Liver Abscess; Abscess; Infections
Keywords: Pyogenic Liver abscess; Liver histological change
MeSH Terms: conditions — Liver Abscess, Pyogenic; Liver Abscess; Abscess; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Take 10ml blood sample for each patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pyogenic liver abscess is one of the most common visceral abscesses, its incidence is increasing worldwide. According to the previous literature, the mortality rate of pyogenic liver abscess is as high as 31% and become a serious social health problem. However, the data of prospective observational real-world studies are scarce and no relevant research of the liver histological change has been reported, so the long-term prognosis and the risk factors for pyogenic liver abscess are still unknown. Patients will be followed up prospectively for a period of 2 years and observed clinical prognosis (all-cause mortality, the recurrence rate, and the rehospitalization rate). The investigators will investigate the predictive value of clinical risk factors for clinical prognosis and establish clinical prediction models to predict the long-term prognosis of pyogenic liver abscesses.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age;
* Irrespective of gender;
* Symptomatic patients of liver abscess confirmed with radiology imaging, either by ultrasonography or computed tomography scan.

Exclusion Criteria:

* Patients <18 years old;
* Pregnancy at presentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years of age admitted for pyogenic liver abscesses
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Proportion and causes of deaths within 2 years of discharge from hospital | 2 years
  Define the proportion and causes of deaths within 2 years of discharge from hospital for patients admitted to the Department for pyogenic liver abscesses.
Proportion and causes of re-hospitalization within 2 years of discharge from hospital | 2 years
  Define the proportion and causes of re-hospitalization within 2 years of discharge from hospital for patients admitted to the Department for pyogenic liver abscesses.

SECONDARY OUTCOMES:
The recurrence rate of pyogenic liver abscess | 2 years
  Development new liver abscess after clinical cure during the 2 years follow up period
The number of participants with Histological Change in the Liver | 2 years
  Assessment of histological change in the liver by using ultrasonography or transient elastography during the 2 years follow up period

CONTACTS AND LOCATIONS:
Locations (1):
- NanFang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers except for those are directly involved with this study.